CLINICAL TRIAL: NCT04653805
Title: Differences of the Cardiovascular Risk Factors Therapeutic Approach in T2DM Population According to Gender
Brief Title: Therapeutic Approach of Cardiovascular Risk Factors in T2DM by Gender
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Other Study IDs: 7Z20/036
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes; Cardiovascular Risk Factor; Gender
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Current clinical practice in primary care of patients with type 2 diabetes mellitus

SUMMARY:
Background: Patients with type 2 diabetes mellitus (T2DM) are at 2- to 4-fold higher risk of cardiovascular mortality compared with non-diabetic subjects. Cardiovascular disease (CVD) is the main cause of death in almost half of diabetic population in Spain. Female patients with T2DM have up to 40% excess risk of CVD compared with men and the causes are still unknown. It is argued that a tight control of cardiovascular risk factors could improve the situation.

Hypothesis: The cardiovascular risk factors management in women with T2DM is different than in men with T2DM.

Aims: To assess the therapeutic approach of cardiovascular risk factors and the occurrence of cardiovascular events among women in comparison to men with T2DM.

Methodology: Observational study based on clinical records of primary health care from T2DM patients in Catalonia (2007-2013).

Source: SIDIAP database. Analysis: The two study groups (women and men) will be matched to ensure balance in terms of basal comorbidities and previous cardiovascular disease in order to describe the study group characteristics and to perform a multivariate modeling approach.

Applicability and Relevance: This study is intended to serve to identify the points of improvement of the cardiovascular risk factors therapeutic approach in women.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients > 30 years of age with a clinical record in the SIDIAP database.
* Patients with a diagnosis of type 2 diabetes (codes ICD10: E11, E11.0-E11.9, E14, E14.0-E14.9) on DTALL-30Jun of each year

Exclusion Criteria:

- Patients with a diagnosis of type 1 diabetes (E10), gestational diabetes (O24), secondary diabetes (E12) or any other type of diabetes (E13)

Ages: 31 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is selected from 5,8 million people from the 282 primary care centres of the Catalan Health Service identified with an anonymized personal identifier and included in a unique patient registry called "SIDIAP" for primary care in Catalonia
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Age | 2007-2013
  Age registered on the date of data extraction (DTALL-30Jun)
Gender | 2007-2013
  Gender registered on the date of data extraction (DTALL-30Jun)
Date of DM diagnosis | 2007-2013
  DM onset date registered on the date of data extraction (DTALL-30Jun)
Diagnosis of the most common cardiovascular risk factors | 2007-2013
  High Blood Pressure (>140/90mm Hg), Dyslipidaemia, Smoking and Obesity
Level of of glycated haemoglobin (HbA1c) | 2007-2013
  The value closer and prior to data extraction (DTALL-30Jun) will be considered and a window of up to a year before the DTALL accepted
Average of the three last measurements of systolic and diastolic blood pressure | 2007-2013
  A window of up to a year before the DTALL date will be accepted. If there are no 3BP measurements, the ones available closer to DTALL will be accepted.
Levels of Total Cholesterol (TC), LDL Cholesterol (LDL-C), HDL Cholesterol (HDL-C) and triglycerides (TGC) | 2007-2013
  A window of up to a year before the DTALL date will be accepted
Body Mass Index (BMI) | 2007-2013
  A window of up to a year before the DTALL-30Jun will be accepted. Height will be measured in m and weight in kg
Kidney function: glomerular filtration estimated by MDRD | 2007-2013
  The value closer and prior to data extraction (DTALL-30Jun) will be considered and a window of up to a year before the DTALL accepted
Kidney function: urinary albumin excretion (albumin/creatinine ratio) | 2007-2013
  The value closer and prior to data extraction (DTALL-30Jun) will be considered and a window of up to a year before the DTALL accepted
Use of hypoglycaemic agents and insulin on the DTALL-30Jun | 2007-2013
  Data of use will be obtained from the pharmacy billing of the Catalan Health Service (CatSalut).
Use of antihypertensive, hypolipidemic, antiplatelet and anticoagulant agents on the DTALL-30Jun | 2007-2013
  Data of use will be obtained from the pharmacy billing of the Catalan Health Service (CatSalut)
Cardiovascular disease registered on the DTALL-30Jun | 2007-2013
  Coronary artery disease, cerebrovascular disease and peripheral artery disease with codes
Causes of mortality in the population with type 2 diabetes during the study period | 2007-2013
  Causes of mortality in the population with type 2 diabetes during the study period
Diagnosis of Diabetic retinopathy | 2007-2013
  Diagnosis of Diabetic retinopathy
Number of visits with the primary care team in the previous 12 months | 2007-2013
  A window of up to a year before the DTALL-30Jun will be considered

CONTACTS AND LOCATIONS:
Overall Officials: Didac Mauricio Puente, MD, PhD, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Anna Ramirez-Morros, RN, Principal Investigator — Institut Català de la Salut
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain